CLINICAL TRIAL: NCT01538953
Title: Pakistan Flocculent Health Outcome Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Health Oriented Preventive Education (Other); Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC3794
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Diarrhea
Keywords: diarrhea; handwashing; point-of-use water treatment; diarrhea longitudinal prevalence
MeSH Terms: conditions — Diarrhea | interventions — Hand Disinfection; Water Purification; Sodium Hypochlorite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Handwashing (Experimental): participants received weekly, in-home handwashing promotion and soap as needed
  Interventions: Other: handwashing
- handwashing and water treatment (Experimental)
  Interventions: Other: handwashing; Other: flocculent-disinfectant for water treatment
- Water treatment with sodium hypochlorite (Experimental)
  Interventions: Other: water treatment with sodium hypochlorite
- Water treatment with flocculent-disinfectant (Experimental): participants received a supply of flocculent-disinfectant product and instruction to use it to treat drinking water
  Interventions: Other: flocculent-disinfectant for water treatment
- Control (No Intervention)

INTERVENTIONS:
Other: handwashing — participants received weekly in-home handwashing promotion and soap as needed
  Arms: Handwashing; handwashing and water treatment
Other: flocculent-disinfectant for water treatment — participants received a supply of flocculent-disinfectant product for water treatment and instruction in how to use it
  Arms: Water treatment with flocculent-disinfectant; handwashing and water treatment
Other: water treatment with sodium hypochlorite — participants received a supply of dilute sodium hypochlorite and instruction to treat drinking water with it
  Arms: Water treatment with sodium hypochlorite

SUMMARY:
This study is designed to evaluate the effect of different methods of drinking water treatment on the occurrence of diarrhea among children living in squatter settlements in Karachi, Pakistan, and the marginal benefit of adding handwashing to water treatment. 260 households will receive a new product which combines flocculation with chlorination to produce clearer, less chemically contaminated drinking water. 260 households will receive dilute sodium hypochlorite, i.e. bleach to treat their water. 260 households will receive soap and encouraged to wash their hands regularly. 260 households will receive both soap and the combination flocculation/chlorination water treatment. 260 households will continue their standard water treatment and handwashing practices. The households will be visited each week for 9 months, and the episodes of diarrhea from each child in the household recorded. The rate of diarrhea between the groups will be compared. At the end of 9 months, households who were part of the standard habits and practice group will receive a water storage vessel and disinfectant.

ELIGIBILITY:
Inclusion Criteria:

* households in study neighborhoods
* contain a child < 5 years old
* have access to water for handwashing

Exclusion Criteria:

* participated in handwashing or drinking water treatment programs with HOPE previously

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8949 (Actual)
Dates: Start 2003-03; Primary Completion 2003-12 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
diarrhea longitudinal prevalence

CONTACTS AND LOCATIONS:
Locations (1):
- Health-Oriented Preventive Education, Karachi, Pakistan

REFERENCES:
- [Result] Luby SP, Agboatwalla M, Painter J, Altaf A, Billhimer W, Keswick B, Hoekstra RM. Combining drinking water treatment and hand washing for diarrhoea prevention, a cluster randomised controlled trial. Trop Med Int Health. 2006 Apr;11(4):479-89. doi: 10.1111/j.1365-3156.2006.01592.x. PMID 16553931
- [Result] Boudier E, Zurlinden B, Cour A, Rognon M, Devalland-Monnin C, Nirhy-Lanto A, el Khadissi H. [Antenatal diagnosis of achondrogenesis. Two successive cases in the same family]. J Gynecol Obstet Biol Reprod (Paris). 1991;20(5):623-6. French. PMID 1955657
- [Derived] Bowen A, Agboatwalla M, Luby S, Tobery T, Ayers T, Hoekstra RM. Association between intensive handwashing promotion and child development in Karachi, Pakistan: a cluster randomized controlled trial. Arch Pediatr Adolesc Med. 2012 Nov;166(11):1037-44. doi: 10.1001/archpediatrics.2012.1181. PMID 22986783